CLINICAL TRIAL: NCT02554097
Title: Optimization and Cost-effective Analysis of Secondary Biliary Stones' Managements - A Multicenter, Prospective and Retrospective Cohort Study Based on Case Register System
Brief Title: Chinese Registry Study on Treatment of Cholecysto-Choledocholithiasis
Acronym: CREST Choles
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking University First Hospital (Other); Xuanwu Hospital, Beijing (Other); Capital Medical University (Other); Peking University Third Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Tongren Hospital (Other); LanZhou University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shanghai Zhongshan Hospital (Other); Peking University (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Doctor, Beijing Friendship Hospital
Other Study IDs: CR-CREST Choles
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Gallstones; Cholelithiasis; Cholecystolithiasis; Choledocholithiasis
Keywords: laparoscopic transcystic common bile duct exploration; laparoscopic common bile duct exploration; endoscopic sphincterotomy,; cost-effective analysis
MeSH Terms: conditions — Gallstones; Cholelithiasis; Cholecystolithiasis; Choledocholithiasis | interventions — Sphincterotomy, Endoscopic; Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- EST+LC group: Patients accept the management of endoscopic sphincterotomy and laparoscopic cholecystectomy.
  Interventions: Procedure: endoscopic sphincterotomy; Procedure: laparoscopic cholecystectomy
- LCBDE+LC group: Patients accept the management of laparoscopic common bile duct exploration and laparoscopic cholecystectomy.
  Interventions: Procedure: laparoscopic common bile duct exploration; Procedure: laparoscopic cholecystectomy
- LTCBDE+LC group: Patients accept the management of laparoscopic transcystic common bile duct exploration and laparoscopic cholecystectomy.
  Interventions: Procedure: laparoscopic transcystic common bile duct exploration; Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: endoscopic sphincterotomy — Sphincterotomy (EST) is performed to remove the common bile duct stone.
  Groups: EST+LC group
Procedure: laparoscopic common bile duct exploration — Transductal exploration was carried out to remove the common bile duct stone. Primary closure or a T tube drainage was performed according to the results of transductal surgery.
  Groups: LCBDE+LC group
Procedure: laparoscopic transcystic common bile duct exploration — A wide local dissection of Calot's triangle is performed and a 2.8mm, 3-mm or 5-mm flexible choledochoscope according to the diameter of the cystic duct is inserted through the cystic duct into the common bile duct. After the common bile duct stone is removed, the cystic duct was ligated with Hem-o-lok.
  Groups: LTCBDE+LC group
Procedure: laparoscopic cholecystectomy — Laparoscopic cholecystectomy is performed to remove the gallbladder.

SUMMARY:
Patients with gallstone and confirmed common bile duct stones are registered in this study. The three managements for common bile duct stones are endoscopic sphincterotomy (EST), laparoscopic common bile duct exploration (LCBDE) and laparoscopic transcystic common bile duct exploration (LTCBDE). Patients will be assessed at baseline, preoperative investigations, operative method, operative time, conversion to open procedure, intraoperative and postoperative complications, and the presence of retained and recurrent stones. All patients were followed up for 3 years by telephone interview ang outpatient visits. Abdominal US and liver function tests were carried out whenever any abdominal symptom appeared during the follow-up period. If there were unusual findings, magnetic resonance cholangiopancreatography(MRCP) was carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 - 80 years.
* Patients diagnosed with gallstones.
* Patients diagnosed with common bile duct stone by one of the three exam (MRI、MRCP and CT).
* Patients diagnosed with common bile duct stone by intro-operative cholangiography or transcystic exploration.
* Patients accepted one of the three managements (EST+LC, LCBDE and LTCBDE).

Exclusion Criteria:

* Combined with Mirizzi syndrome and intrahepatic bile duct stones
* Previous EST/endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic biliary drainage (PTBD)
* History of upper abdominal surgery.
* Serious heart,brain,lung, metabolic diseases history.
* Pregnant women
* Unwillingness or inability to consent for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are diagnosed with gallstones and common bile duct stones.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse outcomes | 3 years
  The patients with complication / the total patients

SECONDARY OUTCOMES:
Incremental cost-effectiveness ratio | 3 years
  the average incremental cost associated with 1 additional unit of the measure of effect
Hospital stay | 3 years
  The total days in hospital
Acute cholangitis rate | 30 days
  The patients with acute cholangitis / the total patients
Bile leakage rate | 30 days
  The patients with bile juice found in the abdominal cavity after procedures / the total patients
Stricture of the bile duct rate rate | 3 years
  The patients with any stricture appeared after the procedures / the total patients
Mortality | 3 years
  Number of death connected with the procedures and complications / total patients
Perforation Rate | 30 days
  The patients with perforation after the procedures / the total patients
Hemorrhage Rate | 3 years
  The patients with hemorrhage after the procedures / the total patients
Operation time | 3 years
  The total time of all the procedures (min)
Acute pancreatitis Rate | 30 days
  The patients with acute pancreatitis after the procedures / the total patients

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Doctor, Study Chair — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhu JG, Wu S, Feng Q, Li F, Han W, Xiu D, Tan H, Fu J, Li X, Shang D, Liu H, Li B, Yang L, Kong Y, Zhan S, Guo W, Zhang ZT. Protocol for the CREST Choles (Chinese REgistry Study on Treatment of Cholecysto-Choledocholithiasis) study: an ambispective, multicenter, observational, open-cohort study. BMJ Open. 2019 Nov 24;9(11):e030293. doi: 10.1136/bmjopen-2019-030293. PMID 31767583